CLINICAL TRIAL: NCT03826914
Title: The Effects of the Dietary Supplement CardioFlex Q10 on Reducing Cardiovascular Disease Risk Factors in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CardioFLex Q10
Record Dates: First submitted 2018-11-29; First posted 2019-02-01 (Actual); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2019-12

CONDITIONS: Cardiovascular Diseases; Cardiovascular Abnormalities; Heart Attack; Stroke; Hypertension
Keywords: dietary supplements; cardiovascular diseases; heart attack; stroke; hypertension; amino acids; electrolytes; antioxidants
MeSH Terms: conditions — Cardiovascular Diseases; Cardiovascular Abnormalities; Myocardial Infarction; Stroke; Hypertension

STUDY DESIGN:
Intervention Model Description: A 90-day double blinded controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The selected participants will be randomly assigned in equal numbers to the experimental or control group. Participants in the experimental group will be given 1 serving (10g) of Cardioflex each day. Participants in the control group will be given a flavored 10g placebo that looks and tastes exactly like Cardioflex. Participants will be instructed to consume the beverage in 500mL of water upon waking each morning, prior to eating or drinking anything else.
  The clinical trial is double blinded so neither the participants or investigators will know which experimental group they are in until the data collection period is over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will be given 1 serving (10g) of Cardioflex each day.
  Interventions: Dietary Supplement: CardioFlex Q10
- Control Group (Placebo Comparator): Participants in the control group will be given a flavoured 10g placebo that looks and tastes exactly like Cardioflex.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CardioFlex Q10 — CardioFlex Q10 is a cardiovascular health supplement developed to increase collagen production, repair connective tissues, and help the body metabolize fats and protein. CardioFlex Q10 contains high amounts of lysine, proline and vitamin C, which the body requires to produce connective tissue (collagen). CardioFlex Q10 also includes additional supporting nutrients such as vitamin E, selenium, bio flavonoids, Coenzyme Q10 (Ubiqionol) and magnesium. The ingredients in CardioFlex Q10 help regulate the body's production of cholesterol, strengthen the arteries and heart, and reverse oxidation.
  Arms: Experimental group
Dietary Supplement: Placebo — Isocaloric maltodextrin placebo that looks and tastes identical to CardioFLex Q10
  Arms: Control Group

SUMMARY:
Cardiovascular diseases (CVD), primarily heart disease and stroke, are the leading causes of death and prescription drug use in Canada. Research on certain dietary supplements looks promising as a way to help reduce CVD risk factors. Studies show that supplementation of certain nutrients such as antioxidants, amino acids, electrolytes, vitamins and minerals may effectively reduce cardiovascular risk factors. The dietary supplement CardioFlex Q10, which is high in the aforementioned components, was developed to help regulate the body's production of cholesterol, strengthen the arteries and heart, and reverse oxidation.

The overall objective of this study is to determine if 90 days of supplementing with CardioFlex Q10 can reduce CVD risk factors in adults, independent of other dietary or physical activity changes.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether or not daily supplementation with the dietary supplement CardioFlex Q10 for 90 days can reduce cardiovascular risk factors in healthy adults. The health markers that will be tested include the participant's waist circumference, body weight, body mass index (BMI), atherosclerosis risk factors (blood pressure, plethysmogram (PTG) wave form, heart rate variability, accelerated plethysmograph (APG) type (biological age of arteries)), and blood work including total plasma lipid profile (total cholesterol (TC), high density lipoprotein (HDL), low density lipoprotein (LDL), triglycerides (TGs)), kidney and liver function (alanine aminotransferase (ALT), aspartate aminotransferase (AST), Lactate dehydrogenase (LDH), Blood Urea Nitrogen (BUN), creatinine), and inflammatory and endothelial function biomarkers (C-reactive protein (CRP), Interleukin-6 (IL-6), soluble intercellular cell adhesion molecule-1 (sICAM-1), soluble vascular cell adhesion molecule-1 (sVCAM-1) ).

All health markers will be tested the day before starting the study and the day after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65
* An accelerated plethysmograph (APG) type (biological age of arteries) of D, E, F or G and/or a high density lipoprotein (HDL) to total cholesterol (TC) ratio of ≤24 percent

Exclusion Criteria:

* Have used prescription cholesterol or blood pressure medication in the last 3 months
* Perform more then 150 minutes of moderate to rigorous activity per week
* Pregnant or planning on getting pregnant during the study period

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Semone Myrie, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myers J. Cardiology patient pages. Exercise and cardiovascular health. Circulation. 2003 Jan 7;107(1):e2-5. doi: 10.1161/01.cir.0000048890.59383.8d. No abstract available. PMID 12515760
- [Background] Nunez-Cordoba JM, Martinez-Gonzalez MA. Antioxidant vitamins and cardiovascular disease. Curr Top Med Chem. 2011;11(14):1861-9. doi: 10.2174/156802611796235143. PMID 21506930
- [Background] Manson JE, Gaziano JM, Jonas MA, Hennekens CH. Antioxidants and cardiovascular disease: a review. J Am Coll Nutr. 1993 Aug;12(4):426-32. doi: 10.1080/07315724.1993.10718332. PMID 8409105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of study participants employed several strategies including email, flyers, and in-person presentations.
Groups:
- Control Group: Participants in the control group will be given a flavoured 10g maltodextrin placebo that looks and tastes exactly like Cardioflex Q10.
  Placebo: Maltodextrin placebo that looks and tastes identical to CardioFLex Q10
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 35 | 34
Completed | 34 | 33
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: 69 participants started the clinical trial, 35 in the Cardioflex group and 34 in the Placebo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 participants (1 in cardioflex group and 1 in placebo group) did not complete the study for personal reasons not related to the study
  Participants
    number analyzed (Participants) | 34 | 33 | 67
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 34 | 33 | 67
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants (1 in cardioflex group and 1 in placebo group) did not complete the study for personal reasons not related to the study
  Participants
    number analyzed (Participants) | 34 | 33 | 67
    Female | 22 | 18 | 40
    Male | 12 | 15 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Total Cholesterol After 90 Days
Description: Total cholesterol is the total amount of cholesterol in the blood. Change = Day 90 score - baseline score.
Time Frame: Baseline and 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Cardioflex Group: Participants were given 1 serving (10g) of Cardioflex each day.
- Placebo Group: Participants in the placebo group were given 10g of a maltodextrin placebo per day
Arm/Group | Cardioflex Group | Placebo Group
Number analyzed (Participants) | 34 | 33
mmol/L | -0.57 (1.06) | -1.09 (1.05)
Statistical Analysis 1: Comparison: Cardioflex Group vs Placebo Group; The primary analysis was conducted using the post-treatment biomarker value, comparing the two groups, and controlling for their baseline values by using analysis of covariance. In this study, the dependent variable was the biomarkers being tested, the controlled independent variable was the treatment given and the uncontrolled variables were the baseline differences between participants; Test type: Superiority; p = 0.042, Anaylsis of Covariance — The threshold of significance was P=0.05; Median Difference (Net) = -0.43, 95% CI 2-sided [-0.846 to -0.015] — Placebo - Cardioflex

2. Secondary Outcome: Heart Rate Variability
Description: Heart rate variability is a measure of the variation in time between each heartbeat. Change = day 90 score - baseline score
Time Frame: Baseline and day 90
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Cardioflex: Participants in the Cardioflex group were given 1 serving (10g) of Cardioflex each day.
- Placebo: Participants in the placebo group were given 10g of a maltodextrin placebo each day.
Arm/Group | Cardioflex | Placebo
Number analyzed (Participants) | 34 | 33
ms | 3.49 (10.86) | -6.27 (10.55)
Statistical Analysis 1: Comparison: Cardioflex vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Anaylsis of Covariance — The threshold of significance was P=0.05; Mean Difference (Final Values) = -6.772, 95% CI 2-sided [-11.2 to -2.24]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the 90 day study period.
Groups:
- Experimental Group: Participants were given one serving (10g) of cardioflex daily for 90 consecutive days.
- Control Group: Participants were given one serving of an isocaloric maltodextrin placebo daily for 90 consecutive days.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03826914/Prot_SAP_ICF_000.pdf